CLINICAL TRIAL: NCT02718352
Title: A Naturalistic Study of Adolescents and Young Adults in Treatment for Opioid Dependence
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 16010 17074
Record Dates: First submitted 2016-02-26; First posted 2016-03-24 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Naturalistic Prospective Cohort — Follow subjects through 1 year of naturalistic buprenorphine treatment

SUMMARY:
Many buprenorphine treatment programs do not have services dedicated to adolescents and young adults. As a precursor to developing and evaluating an adolescent and young adult buprenorphine treatment program at APT Foundation Inc, we propose to conduct a 1 year prospective study of 16 to 25 year old treatment-seeking individuals enrolled in the APT Adolescent and Young Adult Suboxone Program

DETAILED DESCRIPTION:
Participants will consent to in-person assessments and monthly chart reviews. We anticipate that the results from this study will inform the development of future services targeted towards adolescents and young adults with opioid dependence.

ELIGIBILITY:
Inclusion Criteria:

* Ages 16 through 25 at time of induction
* Meet criteria for enrollment in the APT Adolescent and Young Adult Suboxone Program (Opioid Dependence per DSM-V criteria; no contraindications to buprenorphine (concomitant benzodiazepine, alcohol use, sedative use),
* Stable enough to participate in outpatient care/intensive outpatient care for at least 12 weeks;
* Can commit to at least 12 weeks of treatment through the APT Adolescent and Young Adult Suboxone Program
* Are willing to provide locator information for follow-up.
* Are fluent in English and have a 6th grader or higher reading level

Exclusion Criteria:

* Have an untreated bipolar or schizophrenic disorder, or active suicidal ideation
* Are physically dependent on alcohol, benzodiazepines, or other sedatives.
* Are in custody of the Department of Children and Families

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Fifty16 to 25 year old opioid treatment-seeking individuals enrolled in the APT Adolescent and Young Adult Suboxone Program.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Opioid Use Patterns | baseline
  To describe the progression of opioid use among adolescents and young adults participating in buprenorphine treatment, the subjects will fill out time line follow back surveys to describe opioid use patterns.
Opioid Use Patterns | 4 weeks
  To describe the progression of opioid use among adolescents and young adults participating in buprenorphine treatment, the subjects will fill out time line follow back surveys to describe opioid use patterns.
Opioid Use Patterns | 8 weeks
  To describe the progression of opioid use among adolescents and young adults participating in buprenorphine treatment, the subjects will fill out time line follow back surveys to describe opioid use patterns.
Opioid Use Patterns | 12 weeks
  To describe the progression of opioid use among adolescents and young adults participating in buprenorphine treatment, the subjects will fill out time line follow back surveys to describe opioid use patterns.
Opioid Use Patterns | 24 weeks
  To describe the progression of opioid use among adolescents and young adults participating in buprenorphine treatment, the subjects will fill out time line follow back surveys to describe opioid use patterns.
Opioid Use Patterns | 52 weeks
  To describe the progression of opioid use among adolescents and young adults participating in buprenorphine treatment, the subjects will fill out time line follow back surveys to describe opioid use patterns.

SECONDARY OUTCOMES:
Opioid Use Patterns | One year
  Urine drug screen results (opioids (and type if noted) benzodiazepines, marijuana, , cocaine, amphetamines) collected monthly from medical charts.
Cigarette Use Patterns | One year
  To describe the progression of cigarette use among adolescents and young adults participating in buprenorphine treatment, the subjects will fill out time line follow back surveys to describe cigarette use patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Camenga, MD, Principal Investigator — Yale University
Locations (1):
- APT Foundation, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No